CLINICAL TRIAL: NCT01125683
Title: A Phase II, Multi-center, Randomized, Double-blind, Placebo-controlled, Crossover Study to Evaluate the Pharmacodynamic Effect of Single and Multiple Oral Doses of AZD1446/ Placebo and a Single Dose of Donepezil on Quantified Electroencephalography and Event-Related Potentials in Patients With AD
Brief Title: To Evaluate Effects of AZD1446, Placebo and Donepezil in Patients With Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor recruitment.
Sponsor: AstraZeneca (Industry)
Responsible Party: MSD, AstraZeneca
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D1950C00011; 2010-018273-38 (EudraCT Number)
Record Dates: First submitted 2010-05-13; First posted 2010-05-18 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Alzheimer´s Disease
Keywords: Phase II; Alzheimer's disease; EEG; cognition; pharmacodynamic
MeSH Terms: conditions — Alzheimer Disease | interventions — 3-(5-chloro-2-furoyl)-3,7-diazabicyclo(3.3.0)octane; Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): 2,5 mg once daily
  Interventions: Drug: AZD1446
- 2 (Active Comparator): single dose of 5 mg
  Interventions: Drug: Donepezil
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo
- 4 (Experimental): 60 mg once daily
  Interventions: Drug: AZD1446
- 5 (Experimental): 60 mg three times daily
  Interventions: Drug: AZD1446

INTERVENTIONS:
Drug: AZD1446 — Capsule, oral single and multiple dose
  Arms: 1; 4; 5
Drug: Donepezil — Capsule, oral and single dose
  Arms: 2
Drug: Placebo — Capsule, oral and single dose
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate whether treatment with single and multiple oral doses of AZD1446 for 1 week will have effect on Quantified Electroencephalography and Event-Related Potentials in patients with Alzheimers Disease. The total treatment period is 9 weeks, divided into 5 equally long sub-periods of 7 days and 4 wash-out periods of 7 days each.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of probable Alzheimer´s Disease
* Hachinski Ischaemic score < 4
* MSE score 18 to 24

Exclusion Criteria:

* History of any clinically significant disease or dementia other than Alzheimer´s Disease
* Current major depressive disorder or other major psychiatric disorders

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-06; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of single and multiple dosing of AZD1446 and a single dose of donepezil on Quantified electroencephalography (qEEG) and Event-related potentials (ERP) in patients with mild-to-moderate AD. | collected from the time of informed consent is signed, throughout the study. The total study period is 9 weeks, divided into 5 equally long treatment periods of 7 days and 4 wash-out periods of 7 days each.

SECONDARY OUTCOMES:
To measure the relationship between plasma concentration of AZD1446/donepezil and qEEG and ERP. | Information on these will be collected from the time of randomization, throughout the study.
To evaluate the correlation between changes in qEEG/ERP and changes in cognition, if applicable | Information on these will be collected from the time of informed consent is signed, throughout the study.
Safety as measured by Adverse Events, Vital Signs, ECGs, Clinical Chemistry, Haematology, Urinalysis and Physical Examination. | Information on these will be collected from the time of informed consent is signed, throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Märta Segerdahl, MD, PhD, Study Director — AstraZeneca
Locations (7):
- Russia (3):
  - Research Site, Kazan'
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Ukraine (4):
  - Research Site, Kiev, Ukraine
  - Research Site, Dnipropetrovsk
  - Research Site, Luhansk
  - Research Site, Vinnytsia